CLINICAL TRIAL: NCT00460850
Title: An Open Label Study to Evaluate the Effect of PEGASYS on ALT and HBV DNA Levels in Patients With Lamivudine-Resistant HbeAg-Negative Chronic Hepatitis B
Brief Title: A Study of PEGASYS (Peginterferon Alfa-2a (40KD)) in Patients With Lamivudine Resistant HBeAg-Negative Chronic Hepatitis B.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low recruitment rate due to treatment regimen change
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Clinical Trials, Study Director, Hoffmann-La Roche
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML20135
Record Dates: First submitted 2007-04-16; First posted 2007-04-17 (Estimated); Last update posted 2008-06-30 (Estimated); Status verified 2008-06

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — peginterferon alfa-2a

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: peginterferon alfa-2a (40KD) [PEGASYS]

INTERVENTIONS:
Drug: peginterferon alfa-2a (40KD) [PEGASYS] — 180 micrograms sc weekly for 48 weeks

SUMMARY:
This single arm study will evaluate the efficacy and safety of PEGASYS in patients with lamivudine resistant HBeAg negative chronic hepatitis B. Patients will receive PEGASYS 180 micrograms s.c. weekly for 48 weeks; following this, there will be a 48 week period of treatment-free follow-up. The anticipated time on study treatment is 3-12 months, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, 18-65 years of age;
* HBeAg negative chronic hepatitis B;
* treated with lamivudine for >=6 months;
* demonstrated lamivudine resistance;
* compensated liver disease.

Exclusion Criteria:

* severe hepatic dysfunction;
* previous treatment with antivirals other than lamivudine;
* immunosuppressant treatment in past 6 months;
* co-infection with hepatitis A, C, or D virus or human immunodeficiency virus;
* medical condition associated with chronic liver disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-09; Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Normalization of ALT, and HBV-DNA <10,000 copies/mL | Week 96

SECONDARY OUTCOMES:
Normalization of ALT, and HBV-DNA <10,000 copies/mL | Weeks 48 and 72
HBsAg loss and anti-HBs seroconversion | Weeks 48, 72 and 96
AEs and lab parameters | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (4):
- Turkey (Türkiye) (4):
  - Ankara
  - Antalya
  - Istanbul
  - Izmir